CLINICAL TRIAL: NCT00508222
Title: A Pilot, Prospective, Open-label Study to Evaluate the Safety and Efficacy of Kaletra® Monotherapy in HIV/HCV Co-infected Subjects.
Brief Title: Kaletra Monotherapy in HIV/HCV Co-infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007217-01H; A06-321
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: HIV; HCV; HIV/HCV Co-infection; Kaletra Monotherapy; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Kaletra Tablets — Kaletra 800/200 OD

SUMMARY:
The study has been designed to test the hypothesis that in patients co-infected with HIV and HCV who exhibit maximal virologic suppression on a double class antiretroviral (ARV) regimen, including two Nucleoside Reverse Transcriptase Inhibitors (NRTIs) and a Non-nucleoside Reverse Transcriptase Inhibitors (NNRTI) or a Protease Inhibitor (PI) (boosted or not with ritonavir), simplification of highly active antiretroviral therapy (HAART) to Kaletra® monotherapy will represent a viable strategy without any negative impact on the virologic control of HIV infection.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine how safe and effective the drug Kaletra® is in treating HIV when it is administered without any other antiretroviral drugs (monotherapy). Kaletra® is 2 protease inhibitors (lopinavir and ritonavir) combined in one dosage form.

Kaletra monotherapy is experimental and subjects eligible to the study are switching from a successful conventional triple therapy to an unproven experimental therapy.

Approximately 40 HIV/HCV coinfected participants, aged over 18 years will participate in this study.

ELIGIBILITY:
Inclusion Criteria

1. Subject has confirmed his or her willingness to participate in the study after being informed of all aspects of the trial that are relevant to his or her decision to participate, by signing and dating the IRB / IEC approved informed consent form.
2. Subject is both HIV positive and HCV positive (must be viremic for HCV, not just antibody positive).
3. Subject is 18 years of age or older.
4. Subject must have an undetectable viral load (VL) less than 50 copies/ml for the last 6 months on HAART therapy.
5. Subject must not be taking any medication that could interact with Kaletra® to enhance hepatic toxicity.
6. Subject's serum AST and ALT levels must be <5 times normal (grade 2 or less) at the start of the study.
7. Subject must not harbour viral strains that are resistant to Kaletra® at the start of the study.
8. Subject has a Karnofsky Score 70 or greater.
9. If female, subject must have a negative pregnancy test and agree to use, for the duration of the study, a barrier method of birth control that has a history of proven reliability as judged by the investigator.
10. Subject does not require and agrees not to take, for the duration of the study, any medication that is contraindicated with Kaletra® (list will be in the protocol).

Exclusion Criteria

1. Subject has active hepatitis B (HbsAg +).
2. Subject has a history of substance abuse or psychiatric illness that could preclude compliance with the protocol.
3. Subject has any of the following abnormal laboratory test results at screening:

   * Hemoglobin 8.0 g/dL or more
   * Absolute neutrophil count 500 cells/mL or more
   * Platelet count 20,000/mL or more
   * ALT or AST 5x Upper Limit of Normal (ULN) or more
   * Creatinine 1.5 x ULN or more
4. Female subject is pregnant or lactating.
5. Subject has received an investigational drug within 30 days prior to the initiation of study dosing.
6. Subject exhibits viral strains that are resistant to lopinavir.
7. Subject is receiving systemic chemotherapy.
8. The subject, in the opinion of the principal investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-06; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the safety and efficacy of Kaletra® (lopinavir/ritonavir) monotherapy in the treatment of patients co-infected with HIV and HCV. | 48 weeks
  patients on cART switched to Kaletra monotherapy an monitored for 48 weeks thereafter

SECONDARY OUTCOMES:
To investigate and compare the pharmacokinetics (PK) of Kaletra® monotherapy at steady-state between co-infected subjects with advanced liver fibrosis (stage 3-4) and those with minimal liver disease (stage 0-2) | 24 weeks
  PK measured at week 4 and 24
To study compliance of subjects | 48 weeks
  adherence assessed at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Cooper, MD, Principal Investigator — OHRI
Locations (2):
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - The Ottawa Hospital, General Campus, Ottawa, Ontario